CLINICAL TRIAL: NCT04215692
Title: Lung Ultrasound-guided Fluid Therapy in Pediatric Intensive Care Unit Patients
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment goal not met. Lack of personnel to complete the trial.
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Collaborators: Centenario Hospital Miguel Hidalgo (Other)
Responsible Party: Principal Investigator, Juan Manuel Marquez Romero, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2019-R-14
Record Dates: First submitted 2019-12-27; First posted 2020-01-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Fluid Overload Pulmonary Edema; Fluid Overload; Pneumonia, Ventilator-Associated; Fluid Overload Without Edema
Keywords: pediatric intensive care; lenght of stay
MeSH Terms: conditions — Edema; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound Guided Fluid Therapy (Experimental)
  Interventions: Diagnostic Test: Pulmonary ultrasound
- Conventional Fluid Therapy (No Intervention)

INTERVENTIONS:
Diagnostic Test: Pulmonary ultrasound — Pulmonary ultrasound is a basic application of critical ultrasound, defined as a loop associating urgent diagnoses with immediate therapeutic decisions.
  Arms: Ultrasound Guided Fluid Therapy

SUMMARY:
A randomized clinical trial to evaluate the effect of using pulmonary ultrasound to guide fluid therapy on distinct variables.

DETAILED DESCRIPTION:
In this randomized clinical trial, the investigators will evaluate the effect of guiding fluid therapy by pulmonary ultrasound on the following variables:

Length of stay in the pediatric ICU Duration of mechanical ventilation Oxygenation index PaO2/FiO2

ELIGIBILITY:
Inclusion Criteria:

* All pediatric inpatient intensive care unit admissions
* Signed Informed Consent Form

Exclusion Criteria:

* Cyanotic congenital heart disease
* Not requiring mechanical ventilation

Ages: 1 Week to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Length of stay | through study completion, an average of 14 days
  Number of days that the patient requires care in the ICU

SECONDARY OUTCOMES:
Oxygenation Index | Daily through study completion, an average of 14 days
  Measure of the fraction of inspired oxygen (FiO2) and its usage within the body.
PaO2/FIO2 | Daily through study completion, an average of 14 days
  Ratio of arterial oxygen partial pressure to fractional inspired oxygen
Duration of mechanical ventilation | through study completion, an average of 14 days
  Days that a patient remains under mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Centenario Hospital Miguel Hidalgo, Aguascalientes, Aguascalientes, Mexico

IPD SHARING:
Plan to Share IPD: No
We are not planning to share the data.